CLINICAL TRIAL: NCT06961747
Title: An Open-Label, Repeated-Dose Assessment of Zilucoplan Concentration in Breast Milk of Healthy Lactating Women
Brief Title: A Study to Assess Zilucoplan Concentration in Breast Milk of Healthy Lactating Women
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: UCB Biopharma SRL (Industry)
Responsible Party: Sponsor
Organization: UCB Pharma (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: UP0137
Record Dates: First submitted 2025-04-29; First posted 2025-05-08 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Healthy Participants
Keywords: Phase 1; Healthy lactating women; zilucoplan; RA101495
MeSH Terms: interventions — zilucoplan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Zilucoplan (Experimental): Study participants enrolled in this arm will receive daily ZLP injections.
  Interventions: Drug: Zilucoplan

INTERVENTIONS:
Drug: Zilucoplan — Dose formulation: Solution for injection. Route of administration: Subcutaneous injection.
  Other Names: RA101495

SUMMARY:
The purpose of this study is to assess the steady state (SS) concentrations of zilucoplan (ZLP) and its major metabolites in mature breast milk of healthy study participants following injection of repeated once-daily doses of ZLP.

ELIGIBILITY:
Inclusion Criteria:

* Study participant must be minimum 18 years at the time of signing the Informed consent form (ICF)
* Study participant is overtly healthy as determined by medical evaluation including medical history, physical examination, laboratory tests, and cardiac monitoring
* Study participant is lactating and will be at least 6 weeks postpartum on Day 1 of the study
* Study participant has already planned, prior to having knowledge of this study, to cease breast milk feeding (by any means) in relation to her current period of lactation
* Study participant agrees to cease breast milk feeding by Day 1 of the study and to not resume breast milk feeding (by any means and of any infant) or donate breast milk following study end for the remainder of her current period of lactation
* Study participant is up to date with vaccinations against meningococcal bacteria (serogroups A, C, W, Y, and B) at least 2 weeks before the first administration of study medication according to the current (at the time of study participant consent) Advisory Committee on Immunization Practices (ACIP) recommendations for meningococcal vaccinations in patients receiving a complement inhibitor
* Study participant is capable of giving signed informed consent

Exclusion Criteria:

* Study participant has a history or presence of/significant history of or current cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrinological, hematological, or neurological disorders capable of significantly altering the absorption, metabolism, or elimination of drugs; constituting a risk when taking the study medication; or interfering with the interpretation of data
* Study participant has any medical, obstetrical, or psychiatric condition that, in the opinion of the investigator, could jeopardize or would compromise the study participant's ability to participate in this study
* Study participant has alanine aminotransferase (ALT), aspartate aminotransferase (AST), or alkaline phosphatase (ALP) >1.0x upper limit of normal (ULN). Tests that result in ALT, AST, or ALP up to 25 percentage (%) above the exclusion limit may be repeated once for confirmation. This includes rescreening. If the repeat values are below the ULN, the study participant will be considered to not meet the exclusion criteria
* Study participant has bilirubin >1.0xULN (isolated bilirubin <1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35%). For participants with a Baseline result >ULN for total bilirubin, a Baseline diagnosis and/or the cause of any clinically meaningful elevation must be understood and recorded in the eCRF
* Study participant has a history of lymphoma, leukemia, or any malignancy within the past 5 years except for basal cell or squamous epithelial carcinomas of the skin that have been resected with no evidence of metastatic disease for 3 years
* Study participant has current or recent systemic infection within 2 weeks before the first administration of study medication or infection requiring intravenous antibiotics within 4 weeks before the first administration of study medication. Note: Study participants with mastitis at Screening that does not meet the criteria for clinically significant infection may be rescreened after the infection is completely resolved
* Study participant has a prior history of meningococcal disease
* Study participant has presence of hepatitis B surface antigen at Screening or within 3 months prior to dosing
* Study participant has a positive hepatitis C antibody test result at Screening or within 3 months prior to starting study medication
* Study participant has a positive hepatitis C RNA test result at Screening or within 3 months prior to first dose of study medication
* Study participant has a positive prestudy drug and/or alcohol screen
* Study participant has a positive human immunodeficiency virus antibody test at the Screening Visit
* Study participant has a positive syphilis test at the Screening Visit

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 15 (Estimated)
Dates: Start 2025-07-09 (Actual); Primary Completion 2026-07-22 (Estimated); Study Completion 2026-07-22 (Estimated)

PRIMARY OUTCOMES:
Concentrations of zilucoplan and its major metabolites (RA103488 and RA102758) in breast milk during 24 hour steady state (SS) Sampling Period | 30 minutes predose on Day 10 and at prespecified intervals (0 to ≤3, >3 to ≤6, >6 to ≤9, >9 to ≤12, and >12 to ≤24 hours) postdose on Day 10
  Maternal breast milk samples will be collected for measurement of zilucoplan and its major metabolites.

SECONDARY OUTCOMES:
Daily Infant Dosage of zilucoplan and its major metabolites (RA103488 and RA102758) from breast milk over a 24 hour SS Sampling Period | 30 minutes predose on Day 10 and at prespecified intervals (0 to ≤3, >3 to ≤6, >6 to ≤9, >9 to ≤12, and >12 to ≤24 hours) postdose on Day 10
  The estimated daily infant dosage level of zilucoplan from breast milk will be calculated based on the concentration of zilucoplan in mature human breast milk for the Pharmacokinetic Set (PKS).
Occurrence of treatment emergent adverse events (TEAEs) | From Day 1 Visit up to the Safety Follow-Up Visit (Week 8)
  An Adverse event (AE) is any untoward medical occurrence in a patient or clinical study participant, temporally associated with the use of study medication, whether or not considered related to the study medication. TEAEs are adverse events do not present prior to the pharmaceutical product administration or an already present event that worsens either in intensity or frequency.
Estimated Relative Infant Dose of ZLP and its major metabolites (RA103488 and RA102758) from breast milk over a 24 hour SS Sampling Period | 30 minutes predose on Day 10 and at prespecified intervals (0 to ≤3, >3 to ≤6, >6 to ≤9, >9 to ≤12, and >12 to ≤24 hours) postdose on Day 10
  The relative daily infant dosage level of zilucoplan from breast milk will be calculated based on the concentration of zilucoplan in mature human breast milk for the Pharmacokinetic Set (PKS).

CONTACTS AND LOCATIONS:
Overall Officials: UCB Cares, Study Director — 001 844 599 2273
Locations (2):
- United States (2):
  - UP0137 2, San Antonio, Texas
  - UP0137 1, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No
Due to the small sample size in this trial, IPD cannot be adequately anonymized i.e., there is a reasonable likelihood that individual participants could be re-identified. For this reason, data from this trial cannot be shared.